CLINICAL TRIAL: NCT05055128
Title: A Randomized Double-blind, Double Dummy, Active Comparator-controlled Dose-finding Study in Patients With Erosive Esophagitis Due to Gastro-esophageal Reflux Disease (GERD) Los Angeles Grade C or D, and Patients With at Least Partial Symptom Response But Endoscopically Still Unhealed After 8 Weeks History of Standard Treatment Healing Course With Proton-pump Inhibitor (PPI), to Investigate Safety, Tolerability, and Healing Rates After 4 Weeks Treatment of X842 or Lansoprazole, and Symptom Pattern During Subsequent 4 Weeks Treatment With Lansoprazole
Brief Title: A Study in Patients With Erosive Esophagitis to Investigate Safety, Tolerability, and Healing Rates After 4 Weeks Treatment of X842 or Lansoprazole and Symptom Pattern During Subsequent 4 Weeks Treatment With Lansoprazole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cinclus Pharma AG (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CX842A2201; 2020-003319-91 (EudraCT Number)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Erosive Esophagitis
Keywords: Lansoprazole; Los Angeles Grade; Double-blind; Active comparator-controlled; Proton-pump inhibitor; Dose selection
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- X842 25 mg BID (Experimental): Patients will receive 2 tablets (X842 25mg + X842 dummy) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 25 mg + X842 dummy) in the evening during 4-week double-blind treatment. Thereafter, patients will receive 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
  Interventions: Drug: X842; Drug: X842 Dummy; Drug: Lansoprazole; Drug: Lansoprazole Dummy
- X842 50 mg BID (Experimental): Patients will receive 2 tablets (X842 50 mg + X842 dummy) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg + X842 dummy) in the evening during 4-week double-blind treatment. Thereafter, patients will receive 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
  Interventions: Drug: X842; Drug: X842 Dummy; Drug: Lansoprazole; Drug: Lansoprazole Dummy
- X842 75 mg BID (Experimental): Patients will receive 2 tablets (X842 50 mg + X842 25 mg) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg + X842 25 mg) in the evening during 4-week double-blind treatment. Thereafter, patients will receive 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
  Interventions: Drug: X842; Drug: Lansoprazole; Drug: Lansoprazole Dummy
- X842 100 mg BID (Experimental): Patients will receive 2 tablets (X842 50 mg×2) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg×2) in the evening during 4-week double-blind treatment. Thereafter, patients will receive 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
  Interventions: Drug: X842; Drug: Lansoprazole; Drug: Lansoprazole Dummy
- Lansoprazole (Active Comparator): Patients will receive 2 tablets (X842 dummy×2) and 1 capsule (Lansoprazole 30 mg) in the morning, and 2 tablets (X842 dummy×2) in the evening during 4-week double-blind treatment. Thereafter, patients will receive 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
  Interventions: Drug: X842 Dummy; Drug: Lansoprazole

INTERVENTIONS:
Drug: X842 — Patients will receive X842 tablets.
  Arms: X842 100 mg BID; X842 25 mg BID; X842 50 mg BID; X842 75 mg BID
Drug: X842 Dummy — Patients will receive matching placebo tablets for X842.
  Arms: Lansoprazole; X842 25 mg BID; X842 50 mg BID
Drug: Lansoprazole — Patients will receive Lansoprazole capsule.
Drug: Lansoprazole Dummy — Patients will receive matching placebo capsules for Lansoprazole.
  Arms: X842 100 mg BID; X842 25 mg BID; X842 50 mg BID; X842 75 mg BID

SUMMARY:
This study will be conducted in patients with erosive esophagitis due to gastro-esophageal reflux disease (GERD) Los Angeles (LA) grades C or D, and in patients with at least partial symptom response but still endoscopically unhealed (LA grades A or B) after 8 weeks history of standard treatment healing course with PPI, designed to support dose selection for Phase 3 and to investigate safety, tolerability, and healing rates after 4 weeks treatment of X842 or Lansoprazole, and symptom pattern during subsequent 4 weeks treatment with Lansoprazole.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active comparator-controlled study with a parallel-group design including four arms with X842 and one arm with Lansoprazole.

Randomization to one of the treatments with X842 twice daily (BID) 25 mg, 50 mg, 75 mg, 100 mg, or Lansoprazole 30 mg once daily (QD) will be based on a 1:1:1:1:1 scheme.

The duration of each patient's participation in the study, including screening, blind treatment period, and open-label treatment period will be approximately 60 days. The patients will be randomized for 4 weeks of double-blind treatment and will be provided with investigational medicinal product for 35 days.

All patients will have an endoscopic evaluation after 4 weeks of treatment. Following the endoscopic evaluation, all patients will receive subsequent 4 weeks of open-label treatment with Lansoprazole. Repeated symptom evaluation to detect symptom patterns will be assessed during this period.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 18 and ≤ 40 kg/m^2 at screening.
2. Gastro-esophageal reflux disease with endoscopically confirmed esophagitis:

   * LA grade C or D ≤7 days before randomization (with or without historical PPI treatment) or
   * LA grade A or B ≤7 days before randomization and history of treatment with the standard healing course of PPI for minimum of 8 weeks prior to screening and ≤7 days of non-treatment during this period and at least partial symptom response during the minimum of 8 weeks of PPI treatment.
3. Willing and able to comply with all aspects of the protocol (including capsule swallowing, diary completion, etc.).
4. Capable of signing informed consent form.

Exclusion Criteria:

1. History or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disease or disorder.
2. Patients with so-called "alarm features" in symptomatology, like odynophagia, severe dysphagia, bleeding, weight loss, anemia, and blood in stool pointing to a possible malignant disease of the gastrointestinal (GI) tract.
3. Present clinically significant psychiatric diagnosis.
4. History of malignancy of any organ system.
5. Presence of esophageal ulcer, stricture, Barrett´s esophagus or suspected esophagitis secondary to infection, inflammatory disease, ingestion of erosive chemicals or history of any surgical or medical condition which might significantly alter the Gastro-oesophageal reflux disease (GERD) status or the absorption, distribution, metabolism or excretion of drugs.
6. Known severe atrophic gastritis.
7. Any planned major surgery within the duration of the study.
8. History of a positive result for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), antibody to Hepatitis B core antigen (anti-HBcAg), or antibody to Hepatitis C virus (anti-HCV) or presence of these findings on screening.
9. History of long QTc syndrome (e.g. QTc ≥450 ms for males and ≥470 ms for females).
10. Cardiac arrhythmias or any clinically significant abnormalities in the resting 12-lead ECG at the time of screening, as judged by the Investigator.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
12. Current or history of alcohol, drug abuse and/or use of anabolic steroids within 2 years prior to screening.
13. Women who are pregnant or breastfeeding.
14. Patients who have previously participated (completed or withdrawn) in this study CX842A2201.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- Genesis Clinical Research - Tampa, Tampa, Florida, United States
- Bulgaria (16):
  - Medical Center Excelsior, Sofia, Sofia-Grad
  - DCC XIV Sofia, Sofia, Sofia-Grad
  - Medical Centre Asklepii, Dupnitsa
  - Medical Center Medconsult Pleven, Pleven
  - DCC-1 Sliven, Plovdiv
  - MHAT "Kaspela", Plovdiv
  - Medical Center Prolet EOOD, Rousse
  - Diagnostive Consultative Center-1 Sliven, Sliven
  - Medical Center Hera - Gastroenterology office, Sliven
  - 2-nd MHAT, Sofia
  - Medical Center Excelsior, Sofia
  - MHAT "Sveti Ivan Rilski" - Sofia, Sofia
  - Medical Center Hera - Gastroenterology office, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora
  - Medical Center "Biomed 99" Ltd, Vidin
  - Mhat "Hristo Botev", Vratsa
- ResTrial GastroEndo s.r.o., Prague, Czechia
- Georgia (5):
  - LTD"Brothers", Batumi, Adjara
  - A. Aladashvili clinic LLC, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - LTD TSMU and Ingorokva High Medical Technology University Clinic, Tbilisi
  - Emergency Cardiology Center named by acad. G. Chapidze, Tbilisi
- Hungary (4):
  - Bekes Megyei Kozponti Korhaz, Dr.Rethy Pal Tagkorhaz, Békéscsaba, Bekes County
  - Szegedi Tudomanyegyetem Általános Orvostudományi Kar, Szeged, Csongrád megye
  - ClinExpert Kft., Budapest, Pest County
  - Pannonia Maganorvosi Centrum Kft, Budapest
- Poland (8):
  - NZOZ "Centrum Medyczne KERMED", Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Szpital Zakonu Bonifratrow Sw. Jana Bozego w Lodzi, Lodz, Lódzkie
  - Oswiecimskie Centrum Badan Klinicznych Medicome Sp. z o.o., Oświęcim
  - ETG Skierniewice, Skierniewice
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw
  - ETG Zamosc, Zamość
- Zvezdara University Medical Center, Belgrade, Serbia
- Ukraine (4):
  - Oblasna komunalna ustanova "Chernivetska oblasna klinichna likarnia", Chernivtsi, Chernivtsi Oblast
  - KNP "Odeska oblasna klinichna likarnia" Odeskoi oblasnoi rady", Odesa, Odesa Oblast
  - Medychnyi Tsentr TOV "KHELS KLINIK" - viddil Gasrtroenterology, Hepatology and Endocrinology, Vinnytsia, Vinnytsia Oblast
  - KU "6-A miska klinichna likarnia", Zaporizhzhia, Zaporizhzhia Oblast

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paper Alert. Eur J Gastroenterol Hepatol. 2025 Jul 1;37(7):887-890. doi: 10.1097/MEG.0000000000003011. Epub 2025 May 28. PMID 40470733
- [Derived] Sharma P, Vaezi M, Unge P, Andersson K, Larsson K, Popadiyn I, Rosenholm M, Rosztoczy A, Yektaei E, Armstrong D. Clinical Trial: Dose-Finding Study of Linaprazan Glurate, A Novel Potassium-Competitive Acid Blocker, Versus Lansoprazole for the Treatment of Erosive Oesophagitis. Aliment Pharmacol Ther. 2025 May;61(10):1590-1602. doi: 10.1111/apt.70109. Epub 2025 Apr 4. PMID 40183130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 36 centers which included 248 patients across 08 countries. The trial began on 11 Aug 2021 (first patient enrolled) and was completed on 01 Sep 2022 (Last patient completed).
Pre-assignment Details: The pre-treatment assessments were performed during the screening period (Day -7 to Day 0) prior to the first dose preferably. All the study assessments were performed as per the schedule of assessments.
Groups:
- X842 25 mg BID: Patients received 2 tablets (X842 25mg + X842 dummy) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 25 mg + X842 dummy) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
- X842 50 mg BID: Patients received 2 tablets (X842 50 mg + X842 dummy) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg + X842 dummy) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
- X842 75 mg BID: Patients received 2 tablets (X842 50 mg + X842 25 mg) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg + X842 25 mg) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
- X842 100 mg BID: Patients received 2 tablets (X842 50 mg×2) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg×2) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
- Lansoprazole: Patients received 2 tablets (X842 dummy×2) and 1 capsule (Lansoprazole 30 mg) in the morning, and 2 tablets (X842 dummy×2) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
Period: Overall Study
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Started | 51 | 48 | 52 | 47 | 50
Completed | 45 | 45 | 50 | 41 | 47
Not Completed | 6 | 3 | 2 | 6 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 2 | 4 | 2
Not completed — Randomized By Mistake | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all patients who have been randomized and received at least 1 dose of study drug.
Groups:
- X842 25 mg BID: Patients received 2 tablets (X842 25 mg + X842 dummy) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 25 mg + X842 dummy) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole | Total
Number analyzed (Participants) | 51 | 48 | 52 | 47 | 50 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (15.99) | 45.3 (14.11) | 48.7 (14.05) | 54.8 (13.26) | 49.1 (15.41) | 49.3 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 22 | 17 | 20 | 96
  Male | 33 | 29 | 30 | 30 | 30 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 49 | 48 | 50 | 47 | 48 | 242
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 50 | 48 | 52 | 47 | 50 | 247
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Esophageal Mucosa Healing
Description: The healing of erosive esophagitis due to gastro-esophageal reflux disease (GERD) was assessed. It supported the dose selection X842,through the assessment of healing of erosive esophagitis due to GERD based on endoscopic assessment after 4 weeks of treatment. The dose that would lead to having 85% of the patients have esophageal mucosa healing after 4 weeks of treatment. Following the endoscopic evaluation, all patients received subsequent 4 weeks of open-label treatment with lansoprazole. Repeated symptom evaluation was assessed during this period to detect the symptom pattern. Endoscopy evaluation at 4 weeks was based on the level and duration of acid control achieved with X842. Symptom evaluation was assessed using the validated patient-reported outcome (PRO) QOLRAD (Heartburn version) and patient diaries (RESQ-eDiary).
Time Frame: Week 4
Population: The FAS consisted of all patients who had been randomized and received at least 1 dose of study drug. FAS erosive is a subset of FAS consisted of patients who had been classified as erosive (Grade A, B, C or D) as screening according to the central reading or imputed by local reading if missing.
Measure: Count of Participants; unit: Participants
Groups:
- X842 75 mg BID: Patients received 2 tablets (X842 50 mg + X842 25 mg) and 1 capsule (Lansoprazole dummy) in the morning, and 2 tablets (X842 50 mg+ X842 25 mg) in the evening during 4-week double-blind treatment. Thereafter, patients received 1 capsule of Lansoprazole 30 mg QD for 4 weeks.
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 38 | 37 | 41 | 33 | 33
Participants | 28 | 28 | 32 | 18 | 20

2. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: The safety and tolerability of the four dose levels of X842 and Lansoprazole were evaluated, where Lansoprazole served as the active comparator. Here TEAE- Treatment-emergent adverse event, ADR- Adverse drug reaction, SAE- Serious adverse event, and AESI- Adverse events of special interest.
Time Frame: From Screening (Day -7 to Day 0) until Week 8
Population: The safety analysis set consisted of all patients who had been randomized and received at least 1 dose of study drug. Patients were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 51 | 48 | 52 | 47 | 50
Participants
  Any AE | 15 | 10 | 12 | 11 | 10
  Any TEAE | 14 | 10 | 12 | 11 | 10
  Any severe TEAE | 1 | 0 | 0 | 0 | 0
  Any treatment related TEAE (ADR) | 4 | 2 | 0 | 2 | 2
  Any TEAE leading to study discontinuation | 1 | 0 | 0 | 1 | 0
  Any SAE | 1 | 0 | 1 | 0 | 0
  Any Serious TEAE | 1 | 0 | 1 | 0 | 0
  Any treatment emergent AESI | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Heartburn-Free 24-hour Days
Description: Heartburn-free in a 24-hour day was a day where patient reported having no burning feeling or pain behind breast or in center of upper stomach for both morning and evening. Percentage of heartburn-free 24-hour days based on eDiary(Reflux Symptom Questionnaire electronic Diary: RESQ-eDiary) was evaluated. Reflux-related symptom pattern was evaluated during initial 4 weeks of treatment with four dose levels of X842 and with Lansoprazole, and symptom pattern during subsequent additional 4 weeks Lansoprazole treatment in open-label. Modified RESQ-eDiary was validated self-reported questionnaire electronic symptom diary. mRESQ-eD has 3 domains [i.e. Heartburn (min-max: 0-10), Other GERD signs/symptoms (min-max:0-15) and Regurgitations/Reflux (min-max: 0-8)]. Endoscopy followed by lansoprazole administration and symptom evaluation using PRO QOLRAD (Heartburn version) and patient diaries assessed acid control achieved with X842 at 4 weeks.
Time Frame: Weeks 1 and 8
Population: The FAS consisted of all patients who had been randomized and received at least 1 dose of the study drug. Here, the "Number Analyzed" in the table represents the count of patients who were measured and analyzed for the specific Outcome Measure during the given week.
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 48 | 46 | 51 | 46 | 48
Percentage of days
  Week 1 | 27.0 (5.80) | 25.1 (5.91) | 29.2 (5.56) | 26.1 (5.86) | 19.1 (5.68)
  Week 8: number analyzed (Participants) | 31 | 34 | 34 | 29 | 32
  Week 8 | 82.4 (6.59) | 73.8 (6.51) | 78.6 (6.19) | 72.2 (6.78) | 59.2 (6.48)

4. Secondary Outcome: Percentage at Most-mild Heartburn 24-hour Days
Description: Heartburn with at most mild symptoms in a 24-hour day was defined as a day where the patient reported having either no symptoms, very mild symptoms, or mild burning feeling or pain behind the breast or in the center of the upper stomach (score between 0-2) for both morning and evening. Heartburn assessed the severity as per the following scores (0=Did not have, 1=Very mild, 2=Mild, 3=Moderate, 4=Moderately severe, 5=Severe). Here higher scores represent the worst outcome, whereas lower scores represent the better outcome. After endoscopic evaluation, patients received lansoprazole, and symptom evaluation was conducted to detect patterns. Endoscopy evaluation at 4 weeks was based on the level and duration of acid control achieved with X842. Symptom evaluation involved the use of validated PRO QOLRAD (Heartburn version) and patient diaries.
Time Frame: Weeks 1 and 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 48 | 46 | 51 | 46 | 48
Percentage of days
  Week 1 | 75.3 (3.78) | 67.9 (3.85) | 79.4 (3.62) | 69.7 (3.81) | 63.1 (3.70)
  Week 8: number analyzed (Participants) | 31 | 34 | 34 | 29 | 32
  Week 8 | 98.5 (4.34) | 96.5 (4.27) | 95.8 (4.08) | 97.1 (4.46) | 92.2 (4.26)

5. Secondary Outcome: Investigator Assessment of Symptoms by Frequency and Severity
Description: Investigator assessed severity and frequency of patients' heartburn, regurgitation, and dysphagia in 7 days. Assessment included both severity grade (for severity, items were coded: none, mild, moderate, severe where none represented no complaints, severe represented incapacitating symptoms) and frequency (for frequency, a 7-graded Likert scale was used, ranging from none to all of time) of symptoms. Symptoms were scored as follows: none (no complaints), mild (aware of symptom, but easily tolerated), moderate (discomforting symptom, sufficient to cause interference with normal daily activities and/or sleep), severe (incapacitating symptom, with inability to perform normal daily activities and/or sleep). Following endoscopic evaluation, patients received lansoprazole and underwent symptom evaluation using validated PRO QOLRAD (Heartburn version) and patient diaries.Here, for frequency- All of the time and None of the time, and for symptoms- none and severe data has been presented.
Time Frame: Weeks 1 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 50 | 46 | 50 | 45 | 48
Participants
  Week 1 (Dysphagia): Frequency- All of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Dysphagia): Frequency- All of the time | 0 | 2 | 0 | 1 | 0
  Week 1 (Dysphagia): Frequency- None of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Dysphagia): Frequency- None of the time | 14 | 10 | 13 | 13 | 11
  Week 8 (Dysphagia): Frequency- All of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Dysphagia): Frequency- All of the time | 0 | 0 | 0 | 1 | 0
  Week 8 (Dysphagia): Frequency- None of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Dysphagia): Frequency- None of the time | 42 | 37 | 43 | 34 | 40
  Week 1 (Heartburn): Frequency- All of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Heartburn): Frequency- All of the time | 4 | 0 | 3 | 3 | 3
  Week 1 (Heartburn): Frequency- None of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Heartburn): Frequency- None of the time | 1 | 0 | 4 | 4 | 1
  Week 8 (Heartburn): Frequency- All of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Heartburn): Frequency- All of the time | 0 | 0 | 0 | 0 | 0
  Week 8 (Heartburn): Frequency- None of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Heartburn): Frequency- None of the time | 38 | 37 | 43 | 33 | 36
  Week 1 (Regurgitation/Reflux): Frequency- All of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Regurgitation/Reflux): Frequency- All of the time | 1 | 0 | 2 | 1 | 0
  Week 1 (Regurgitation/Reflux): Frequency- None of the time: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Regurgitation/Reflux): Frequency- None of the time | 1 | 2 | 4 | 4 | 3
  Week 8 (Regurgitation/Reflux): Frequency- All of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Regurgitation/Reflux): Frequency- All of the time | 0 | 0 | 0 | 1 | 0
  Week 8 (Regurgitation/Reflux): Frequency- None of the time: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Regurgitation/Reflux): Frequency- None of the time | 41 | 36 | 41 | 32 | 39
  Week 1 (Dysphagia): Symptom- None: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Dysphagia): Symptom- None | 14 | 12 | 13 | 15 | 12
  Week 1 (Dysphagia): Symptom- Severe: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Dysphagia): Symptom- Severe | 1 | 2 | 2 | 2 | 1
  Week 8 (Dysphagia): Symptom- None: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Dysphagia): Symptom- None | 42 | 37 | 43 | 35 | 41
  Week 8 (Dysphagia): Symptom- Severe: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Dysphagia): Symptom- Severe | 0 | 0 | 0 | 0 | 0
  Week 1 (Heartburn): Symptom- None: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Heartburn): Symptom- None | 1 | 0 | 4 | 5 | 1
  Week 1 (Heartburn): Symptom- Severe: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Heartburn): Symptom- Severe | 5 | 1 | 4 | 2 | 3
  Week 8 (Heartburn): Symptom- None: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Heartburn): Symptom- None | 38 | 37 | 44 | 33 | 38
  Week 8 (Heartburn): Symptom- Severe: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Heartburn): Symptom- Severe | 1 | 0 | 1 | 0 | 0
  Week 1 (Regurgitation/Reflux): Symptom- None: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Regurgitation/Reflux): Symptom- None | 1 | 3 | 6 | 5 | 3
  Week 1 (Regurgitation/Reflux): Symptom- Severe: number analyzed (Participants) | 50 | 46 | 50 | 45 | 47
  Week 1 (Regurgitation/Reflux): Symptom- Severe | 3 | 3 | 5 | 4 | 2
  Week 8 (Regurgitation/Reflux): Symptom- None: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Regurgitation/Reflux): Symptom- None | 41 | 36 | 41 | 33 | 41
  Week 8 (Regurgitation/Reflux): Symptom- Severe: number analyzed (Participants) | 48 | 46 | 50 | 42 | 48
  Week 8 (Regurgitation/Reflux): Symptom- Severe | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Change From Baseline in Quality of Life in Reflux and Dyspepsia (QOLRAD) Score
Description: Reflux-related symptom pattern was evaluated during initial 4 weeks of treatment with 4 dose levels of X842 and with Lansoprazole, and symptom pattern during subsequent additional 4 weeks of open-label treatment with Lansoprazole. Heartburn version of QOLRAD is a disease-specific instrument containing 25 questions addressing concerns associated with gastrointestinal symptoms. Questions were rated on a seven-grade (1-7) Likert scale, where a score of 1 represented low quality of life, and as score increased, the patient's condition was considered better. Questions were categorized into 5 domains: emotional distress, sleep disturbance, vitality, food/drink problems, and physical/social functioning. The score in each domain was calculated as the mean of all items in that domain. The score ranges from 1 to 175, higher scores mean a better outcome. After endoscopic evaluation, patients received lansoprazole and underwent symptom evaluation using validated PRO QOLRAD and patient diaries.
Time Frame: Baseline, Weeks 1, and 8
Population: The FAS consisted of all patients who had been randomized and received at least 1 dose of study drug. Here, the "Number Analyzed" in the table represents the count of patients who were measured and analyzed for the specific Outcome Measure during the given week.
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
Number analyzed (Participants) | 40 | 40 | 41 | 34 | 41
Scores on scale
  Week 1: Emotional Distress Score | 1.69 (0.247) | 1.55 (0.251) | 1.14 (0.233) | 1.54 (0.255) | 1.34 (0.241)
  Week 8: Emotional Distress Score: number analyzed (Participants) | 27 | 24 | 27 | 22 | 23
  Week 8: Emotional Distress Score | 2.76 (0.265) | 2.51 (0.275) | 1.84 (0.253) | 2.00 (0.278) | 2.19 (0.269)
  Week 1: Food/Drink Problems Score | 1.84 (0.229) | 1.62 (0.232) | 1.32 (0.217) | 1.65 (0.238) | 1.40 (0.223)
  Week 8: Food/Drink Problems Score: number analyzed (Participants) | 27 | 24 | 27 | 22 | 23
  Week 8: Food/Drink Problems Score | 3.08 (0.249) | 2.97 (0.259) | 2.34 (0.240) | 2.28 (0.264) | 2.56 (0.256)
  Week 1: Physical/Social Functioning Score | 1.26 (0.247) | 1.32 (0.252) | 1.02 (0.233) | 1.19 (0.255) | 0.97 (0.241)
  Week 8: Physical/Social Functioning Score: number analyzed (Participants) | 27 | 24 | 27 | 22 | 23
  Week 8: Physical/Social Functioning Score | 2.06 (0.262) | 2.26 (0.271) | 1.57 (0.249) | 1.60 (0.274) | 1.71 (0.265)
  Week 1: Sleep Disturbance Score | 1.60 (0.250) | 1.45 (0.255) | 1.08 (0.236) | 1.49 (0.258) | 1.54 (0.244)
  Week 8: Sleep Disturbance Score: number analyzed (Participants) | 27 | 24 | 27 | 22 | 23
  Week 8: Sleep Disturbance Score | 2.78 (0.266) | 2.48 (0.276) | 1.89 (0.254) | 1.91 (0.279) | 2.37 (0.270)
  Week 1:Vitality Score | 1.55 (0.237) | 1.51 (0.240) | 1.42 (0.224) | 1.50 (0.246) | 1.21 (0.231)
  Week 8: Vitality Score: number analyzed (Participants) | 27 | 24 | 27 | 22 | 23
  Week 8: Vitality Score | 2.84 (0.257) | 2.79 (0.268) | 2.25 (0.247) | 2.21 (0.272) | 2.19 (0.264)

ADVERSE EVENTS:
Time Frame: From Screening (Day -7 to Day 0) until Week 8
Arm/Group | X842 25 mg BID | X842 50 mg BID | X842 75 mg BID | X842 100 mg BID | Lansoprazole
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48 | 0/52 | 0/47 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/48 | 1/52 | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 14/51 | 10/48 | 12/52 | 11/47 | 10/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X842 25 mg BID (N=51) | X842 50 mg BID (N=48) | X842 75 mg BID (N=52) | X842 100 mg BID (N=47) | Lansoprazole (N=50)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X842 25 mg BID (N=51) | X842 50 mg BID (N=48) | X842 75 mg BID (N=52) | X842 100 mg BID (N=47) | Lansoprazole (N=50)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains confidential information about Cinclus Pharma Holding AB. Except as may be otherwise agreed to in writing, by accepting or reviewing these materials, you agree to hold such information in confidence and not to disclose it to others (except where required by applicable law), nor use it for unauthorized purposes. In the event of an actual or suspected breach of this obligation, Cinclus Pharma Holding AB should be promptly notified.

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT05055128/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT05055128/SAP_001.pdf